CLINICAL TRIAL: NCT06535425
Title: Effects of Platelet-Rich Plasma Combined With Isometric Contractions of Quadriceps on Symptoms, Postural Control, Mobility and Inflammatory Markers in Participants With Knee Osteoarthrosis
Brief Title: Participants With Knee Osteoarthrosis
Acronym: KOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Cheng Liang, Principal Investigator, Chengdu Sport University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2022]14; 2024NSFSC0681 (Other Grant/Funding Number: Natural Science Foundation of Sichuan Province)
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthrosis
Keywords: Knee Osteoarthrosis; Platelet-Rich Plasma; Isometric Contractions of Quadriceps
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): Initial Health Education for Participants Initially, all participants received identical health education in the form of thematic lectures once per week for 40 minutes each. The content included the following aspects: emphasising the importance of close cooperation with physicians as key to maintaining health; the process of the occurrence and development of KOA, along with its treatment methods; the role of family and social support in improving the condition; establishing a reasonable daily activity routine, such as protecting the affected knee joint, avoiding long-distance fatigue, mountain climbing, ascending and descending high-rise stairs and various adverse body postures (prolonged standing, kneeling and squatting); and advising those who are overweight to reduce their body weight. On this foundation, the four groups of participants underwent the following interventions.
  Interventions: Other: Control
- Platelet-Rich Plasma (Experimental): The PG and JG were injected with autologous PRP at baseline. The injection was performed by the same clinician with 10 years of experience in knee joint injections. Participants were seated with their knees extended, and the needle was inserted through the joint space into the intra-articular cavity of the knee, administering approximately 2.5 mL of PRP into each knee joint. Thirty millilitres of venous blood were drawn from the participant's elbow vein, and approximately 5 mL of PRP was obtained for bilateral knee joint injection by using a TD5A tabletop low-speed centrifuge manufactured in China. The first centrifugation was performed at 2500 revolutions per minute (rpm) for 3 minutes, followed by a second centrifugation at 2300 rpm for 6 minutes.
  Interventions: Other: Platelet-Rich Plasma; Other: Control
- Isometric Contractions of Quadriceps (Experimental): The IG and JG exercises followed the methods of our previous research, with participants undergoing an 16-week ICQ intervention five times per week. Each session consisted of isometric contractions and relaxations of the quadriceps muscle for 5 seconds each, in sets of 30 repetitions, for a total of 10 sets, with a 30-second rest between sets. During this period, researchers conducted weekly follow-up calls or face-to-face interviews with participants to understand their living conditions, ensuring that they did not change their original lifestyle habits and did not engage in any other form of regular fitness activities. Participants who did not comply were not included in the final data analysis.
  Interventions: Other: Isometric Contractions of Quadriceps; Other: Control
- Platelet-Rich Plasma Combined with Isometric Contractions of Quadriceps (Experimental): Platelet-Rich Plasma Combined with Isometric Contractions of Quadriceps
  Interventions: Other: Platelet-Rich Plasma; Other: Isometric Contractions of Quadriceps; Other: Platelet-Rich Plasma Combined with Isometric Contractions of Quadriceps; Other: Control

INTERVENTIONS:
Other: Platelet-Rich Plasma — The PG and JG were injected with autologous PRP at baseline. The injection was performed by the same clinician with 10 years of experience in knee joint injections. Participants were seated with their knees extended, and the needle was inserted through the joint space into the intra-articular cavity of the knee, administering approximately 2.5 mL of PRP into each knee joint. Thirty millilitres of venous blood were drawn from the participant's elbow vein, and approximately 5 mL of PRP was obtained for bilateral knee joint injection by using a TD5A tabletop low-speed centrifuge manufactured in China. The first centrifugation was performed at 2500 revolutions per minute (rpm) for 3 minutes, followed by a second centrifugation at 2300 rpm for 6 minutes.
  Arms: Platelet-Rich Plasma; Platelet-Rich Plasma Combined with Isometric Contractions of Quadriceps
Other: Isometric Contractions of Quadriceps — The IG and JG exercises followed the methods of our previous research, with participants undergoing an 16-week ICQ intervention five times per week. Each session consisted of isometric contractions and relaxations of the quadriceps muscle for 5 seconds each, in sets of 30 repetitions, for a total of 10 sets, with a 30-second rest between sets. During this period, researchers conducted weekly follow-up calls or face-to-face interviews with participants to understand their living conditions, ensuring that they did not change their original lifestyle habits and did not engage in any other form of regular fitness activities. Participants who did not comply were not included in the final data analysis.
  Arms: Isometric Contractions of Quadriceps; Platelet-Rich Plasma Combined with Isometric Contractions of Quadriceps
Other: Platelet-Rich Plasma Combined with Isometric Contractions of Quadriceps — Platelet-Rich Plasma Combined with Isometric Contractions of Quadriceps
  Arms: Platelet-Rich Plasma Combined with Isometric Contractions of Quadriceps
Other: Control — Initially, all participants received identical health education in the form of thematic lectures once per week for 40 minutes each. The content included the following aspects: emphasising the importance of close cooperation with physicians as key to maintaining health; the process of the occurrence and development of KOA, along with its treatment methods; the role of family and social support in improving the condition; establishing a reasonable daily activity routine, such as protecting the affected knee joint, avoiding long-distance fatigue, mountain climbing, ascending and descending high-rise stairs and various adverse body postures (prolonged standing, kneeling and squatting); and advising those who are overweight to reduce their body weight. On this foundation, the four groups of participants underwent the following interventions.

SUMMARY:
Title: Efficacy and Safety Trial of PRP and ICQ for Elderly Women with KOA

Goal:

To assess if PRP and ICQ reduce symptoms and improve mobility in elderly women with knee osteoarthritis.

Key Questions:

Does PRP and ICQ decrease symptom severity as measured by WOMAC? What side effects occur from PRP and ICQ intervention?

Participants:

Elderly women, aged 60-70, with KOA.

Intervention:

PRP injection and ICQ exercises for 16 weeks.

Procedure:

Daily PRP or placebo for 4 months. Bi-weekly clinic visits for assessments. Weekly health education and lifestyle monitoring.

Measurements:

WOMAC scores, physical mobility tests, and serum biomarkers before and after intervention.

Ethics:

Approved by Chengdu Sport University's Ethics Committee.

Sample Size:

80 participants needed.

Randomization:

Random assignment to PRP, ICQ, or control groups.

This trial aims to determine the benefits and risks of PRP and ICQ in treating KOA in elderly women.

DETAILED DESCRIPTION:
Clinical Trial on the Efficacy and Safety of Platelet-Rich Plasma (PRP) and Isometric Contraction Quadriceps (ICQ) Intervention in Elderly Female Patients with Knee Osteoarthritis (KOA)

Objective:

The primary objective of this clinical trial is to evaluate the effectiveness and safety of Platelet-Rich Plasma (PRP) combined with Isometric Contraction Quadriceps (ICQ) intervention in treating knee osteoarthritis in elderly female patients. The study aims to answer the following questions:

Does the combination of PRP and ICQ reduce the severity of KOA symptoms as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)? What are the potential side effects or complications associated with the PRP and ICQ intervention in elderly patients?

Study Design:

The trial will be a randomized controlled trial comparing the effects of PRP and ICQ intervention with those of a control group. Participants will be randomly assigned to one of four groups: PRP group, ICQ group, joint group (receiving both PRP and ICQ), or control group.

Participants:

Elderly female patients diagnosed with KOA, aged between 60 and 70 years, will be recruited from the Sichuan Provincial People's Hospital. The inclusion and exclusion criteria will be strictly followed to ensure the homogeneity and reliability of the study population.

Intervention:

Participants in the PRP and joint groups will receive an injection of autologous PRP at baseline. The PRP will be prepared from venous blood using a low-speed centrifuge. Participants in the ICQ and joint groups will undergo a 16-week ICQ intervention, performing isometric contractions and relaxations of the quadriceps muscle five times per week.

Procedure:

Participants will receive either PRP injection or a placebo (for the control group) at baseline.

They will undergo a 16-week ICQ intervention if assigned to the ICQ or joint group.

Participants will be required to attend weekly health education sessions for the first month.

They will be followed up weekly through calls or interviews to monitor their adherence to the intervention and to ensure they maintain their usual lifestyle habits.

Assessment:

KOA symptoms will be evaluated using the WOMAC index at baseline and at the end of the 16th week.

Physical mobility will be assessed using the 6-minute walk test (6MWT), time up and go test (TUG), and time up and down stairs (TUDS) at baseline and at the end of the intervention.

Serum levels of inflammation markers and matrix metalloproteinases-13 (MMP-13) will be measured at baseline and post-intervention.

Outcome Measures:

Primary outcomes will include changes in WOMAC scores and physical mobility tests.

Secondary outcomes will include serum levels of TNF-α, IL-1β, and MMP-13.

Ethical Considerations:

The study is approved by the Human Ethics Committee of Chengdu Sport University, and informed consent will be obtained from all participants. The study will adhere to the Declaration of Helsinki.

Sample Size Calculation:

Based on a 4 (group) × 3 (measurement occasions) design, with an estimated dropout rate of approximately 15%, an effect size of 0.3, a power of 0.8, and a significance level of 0.05, a minimum sample size of 80 participants is determined to be necessary.

Randomization:

A total of 92 participants will be recruited and randomly assigned to the four groups using a digital randomization method.

Data Analysis:

Data will be analyzed using appropriate statistical methods to compare the outcomes between the intervention and control groups, as well as among the different intervention groups.

This clinical trial aims to provide evidence-based insights into the efficacy and safety of PRP and ICQ interventions in managing KOA in elderly female patients.

ELIGIBILITY:
Inclusion criteria:

* Female aged between 60 and 70 years
* Participants with KOA severity grades I, II and III were selected
* the study complied with the Declaration of Helsinki, and informed consent was obtained from all participants

Exclusion criteria:

* Need for surgery or pharmacological treatment in the near future
* The presence of neuromuscular diseases and participation in other regular exercise programmes.

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
KOA Symptom Assessment | 16 Weeks
  Symptoms of KOA participants were evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). These questions included assessments of pain (5 questions), stiffness (2 questions) and physical function (17 questions), totalling 24 questions. A 0-100 mm visual analogue scale was used for scoring, which was measured and recorded by a professional by using a ruler. The scores for pain (maximum 500), stiffness (maximum 200) and physical function (maximum 1700) were based on the measured values, with higher scores indicating greater severity.
Balance Ability Testing | 16 Weeks
  The static and dynamic balance of all participants was tested using a BioDex Balance System (BioDex Medical Systems, USA). The test session required participants to stand with both feet, with their hands placed on their sides. The static balance tests included firm surface with eyes closed (FiEC), foam surface with eyes open (FoEO) and foam surface with eyes closed (FoEC) tests.
Isokinetic Muscle Strength Testing of the Knee | 16 Weeks
  The isokinetic strength of both knees (60°/s for 5 repetitions and 180°/s for 5 repetitions) was tested in all participants by using a Germany-manufactured IsoMed 2000 isokinetic testing device. The knee was positioned in a sitting posture with a range of motion of 80°. Participants were required to warm their lower limbs for 10 minutes before the test. The testers provided verbal encouragement throughout the process to ensure reliable test data. The index was the peak torque.
Knee Proprioception Testing | 16 Weeks
  After completing the isokinetic muscle strength test while maintaining the test posture, proprioceptive testing was conducted on the dominant side. The angular velocity was set at 1°/s. The isokinetic device's actuator automatically moved to preset angles of 30° and 60° of knee flexion (with the fully extended knee position at 0°). After each movement to an angle, the actuator returned to the starting position, the participant actively moved to the designated position (the movement stopped automatically after pressing a button), and the difference between the actual and preset angles was recorded. Smaller differences indicate better proprioception, and the average of three trials for each angle was taken.
6-minute walk test | 16 Weeks
  Participants walked back and forth on an outdoor closed corridor (50 m) for 6 minutes, allowing them to slow down or rest if necessary but encouraged to continue walking as much as possible. The time was announced every minute, and the participants were informed of the remaining time 15 seconds before the end of 6 minutes. When the time ended, the participants stopped where they were and marked their position. The total distance walked by the participants was measured in meters.
Time up and go test | 16 Weeks
  Participants sat on a chair with armrests and a backrest (seat height 45 cm, armrest height 20 cm), leaning their backs with their hands on the armrests. A mark was placed 3 meters away from the seat. Upon hearing the 'start' command, participants were required to stand up from the chair, walk forward 3 meters to the mark, turn around and quickly walk back to the chair, then turn and sit down, leaning back against the chair. The time taken from when the participant's back left the chair until they sat down again was recorded in seconds. Participants could practice one or two times before the formal test, which was conducted three times with a 1- to 2-minute interval between each test. The average of the three trials was taken.
Time up and down stairs | 16 Weeks
  Participants were asked to ascend and descend 12 times as quickly as possible, with each step being 18 cm in height and 30 cm in width. Participants could use the handrails during the process. The time required was recorded in seconds using a stopwatch.
TNF-α Testing | 16 Weeks
  Fasting venous blood (5 mL) was collected from all participants upon waking in the morning and centrifuged for 5 minutes (at a centrifugation speed of 3500 r/min and a centrifugation radius of 15 cm) to separate the serum, which was then stored at -80 °C until analysis. The expression levels of serum tumour necrosis factor-α (TNF-α).
IL-1β Testing | 16 Weeks
  Fasting venous blood (5 mL) was collected from all participants upon waking in the morning and centrifuged for 5 minutes (at a centrifugation speed of 3500 r/min and a centrifugation radius of 15 cm) to separate the serum, which was then stored at -80 °C until analysis. The expression levels of serum interleukin-1β (IL-1β) .
MMP-13 Testing | 16 Weeks
  Fasting venous blood (5 mL) was collected from all participants upon waking in the morning and centrifuged for 5 minutes (at a centrifugation speed of 3500 r/min and a centrifugation radius of 15 cm) to separate the serum, which was then stored at -80 °C until analysis. The expression levels of serum matrix metalloproteinases-13.

CONTACTS AND LOCATIONS:
Overall Officials: Yajun Tan, Dr, Principal Investigator — Chengdu Sport University
Locations (1):
- Chengdu Sport University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No